CLINICAL TRIAL: NCT04957719
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of Self-administered Subcutaneous Selatogrel for Prevention of All-cause Death and Treatment of Acute Myocardial Infarction in Subjects With a Recent History of Acute Myocardial Infarction
Brief Title: Selatogrel Outcome Study in Suspected Acute Myocardial Infarction
Acronym: SOS-AMI
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: Viatris Innovation GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID-076A301; 2023-505438-85-00 (EU CTIS Number); 2020-000983-41 (EudraCT Number)
Record Dates: First submitted 2021-06-28; First posted 2021-07-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-04

CONDITIONS: Acute Myocardial Infarction
Keywords: Platelet Aggregation Inhibitors
MeSH Terms: interventions — selatogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Selatogrel (Experimental): Study treatment administration may occur at any time between the randomization visit and the final study visit when the participant experiences symptoms suggestive of an acute myocardial infarction. Study treatment administration triggers protocol pre-defined assessments or visits.
  Interventions: Combination Product: Selatogrel
- Placebo (Placebo Comparator): Study treatment administration may occur at any time between the randomization visit and the final study visit when the participant experiences symptoms suggestive of an acute myocardial infarction. Study treatment administration triggers protocol pre-defined assessments or visits.
  Interventions: Combination Product: Placebo

INTERVENTIONS:
Combination Product: Selatogrel — Selatogrel is a reversible P2Y12 receptor antagonist for subcutaneous administration. Selatogrel will be administered as a liquid formulation in a sealed prefilled syringe in an autoinjector forming an integral ready-to-use, single-dose drug delivery system.
  Participants will self-administer 16 mg of selatogrel subcutaneously with the autoinjector upon occurrence of symptoms suggestive of an acute myocardial infarction. Self-administration encompasses the use of the autoinjector by another person (e.g., partner, close relative, friend, caregiver) who may be called for help during the emergency situation of a suspected AMI.
  Other Names: ACT-246475
  Arms: Selatogrel
Combination Product: Placebo — Placebo will be administered as a liquid formulation in a sealed prefilled syringe in an autoinjector forming an integral ready-to-use, single-dose drug delivery system.
  Participants will self-administer placebo subcutaneously with the autoinjector upon occurrence of symptoms suggestive of an acute myocardial infarction. Self-administration encompasses the use of the autoinjector by another person (e.g., partner, close relative, friend, caregiver) who may be called for help during the emergency situation of a suspected AMI.
  Arms: Placebo

SUMMARY:
This study will randomize patients recently discharged from the hospital with a confirmed diagnosis of type 1 acute myocardial infarction (Thygesen et al. 2018) and having additional cardiovascular risk factors.

DETAILED DESCRIPTION:
The purpose of this study is to assess the clinical efficacy of selatogrel when self-administered upon occurrence of symptoms suggestive of an acute myocardial infarction (AMI) in participants at risk of having a recurrent AMI.

ELIGIBILITY:
Main Inclusion Criteria:

* Confirmed diagnosis of symptomatic type 1 acute myocardial infarction (AMI) ST-Elevation Myocardial Infarction (STEMI) or Non-ST-Elevation Myocardial Infarction (NSTEMI), no longer than 4 weeks prior to randomization.
* Diagnosis of multivessel coronary artery disease defined as ≥ 50% stenosis on 2 or more coronary artery territories, including the left main artery, during a prior cardiac catheterization or cardiac catheterization during the qualifying AMI event and presence of at least 1 of the following risk factors:

  * Second prior AMI,
  * Diabetes mellitus defined by ongoing glucose lowering treatment,
  * Chronic kidney disease defined as estimated glomerular filtration rate less than 60 mL/min/1.73 m2 and either known history of chronic kidney disease or a biomarker of chronic kidney damage,
  * Peripheral artery disease at any time prior to randomization,
  * Absence of, or unsuccessful coronary revascularization of the qualifying AMI.
* Successful self-administered placebo according to the autoinjector instruction for use training during screening.

Main Exclusion Criteria:

* Increased risk of serious bleeding including any of the following:

  * History of intracranial bleed at any time.
  * Known uncorrected intracranial vascular abnormality.
  * Gastrointestinal bleed requiring hospitalization or transfusion within 1 year prior to screening.
  * Already on oral triple antithrombotic therapy (i.e., Dual antiplatelet therapy and oral anticoagulant).
  * Known liver impairment significantly affecting the hepatic function.
  * Current dialysis.
  * Ischemic stroke or transient ischemic attack within 3 months of screening.
* Chronic anemia with hemoglobin < 10 g/dL.
* Chronic thrombocytopenia with platelet count < 100,000/mm3.
* Known hypersensitivity to selatogrel, any of its excipients, or drugs of the P2Y12 class.
* Previous exposure to an investigational drug within 3 months prior to randomization.
* Participation in another clinical trial with an investigational product or device within 3 months prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14000 (Estimated)
Dates: Start 2021-08-14 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Clinical status as assessed by a 6-point ordinal scale | Total duration: up to 7 days
  The clinical status will be assessed using a 6-point ordinal scale after any study treatment self-administration. Only the worst clinical outcome will be retained as the primary efficacy outcome. The 6 mutually exclusive outcomes ranked from worst to best are:
  1. Death (all causes), within 7 days after study treatment administration.
  2. Acute myocardial infarction with compromised electro-hemodynamics, within 2 days after study treatment administration.
  3. ST-Elevation Myocardial Infarction (STEMI), within 2 days after study treatment administration.
  4. High-risk Non-ST-Elevation Myocardial Infarction (NSTEMI), within 2 days after study treatment administration.
  5. NSTEMI with peak cardiac troponin greater than 10 times upper limit of normal, within 2 days after study drug administration.
  6. None of the above
Occurrence of Type 3 or 5 treatment-emergent bleeding events according to the Bleeding Academic Research Consortium (BARC) definition | Total duration: up to 2 days
  The number of:
  * Type 3 treatment-emergent bleeding events and
  * Type 5 treatment-emergent bleeding events
  will be assessed according to the Bleeding Academic Research Consortium (BARC) definition (Mehran et al. 2011), within 2 days after study treatment administration.
  The Bleeding Academic Research Consortium (BARC) definitions are:
  * Type 3, bleeding is divided into 3 categories, a through c, and includes clinical, laboratory, and/or imaging evidence of bleeding with specific healthcare provider responses.
  * Type 5, bleeding is fatal.

SECONDARY OUTCOMES:
Occurrence of death, non-fatal acute myocardial infarction, hospitalization or unplanned emergency department visit for heart failure (Composite endpoint) | Total duration: up to 30 days
  Occurrence death, non-fatal acute myocardial infarction, hospitalization or unplanned emergency department visit for heart failure within 30 days after any self-administration.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Viatris Innovation GmbH
Locations (700):
- United States (82):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - Birmingham VA Health Care System, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cardiovascular Associates of the Southeast, Birmingham, Alabama
  - Grandview Medical Center and Affinity Cardiovascular Specialists, LCC, Birmingham, Alabama
  - Heart Center Research, LLC, Huntsville, Alabama
  - Dignity Health Mercy Gilbert Medical Center, Gilbert, Arizona
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of Arizona - Sarver Heart Center, Tucson, Arizona
  - Northeast Arkansas Charitable Foundation, Inc.- NEA Baptist Clinic, Jonesboro, Arkansas
  - Amicis Research Center., Anaheim, California
  - John Muir Health, Concord, California
  - Long Beach VA Healthcare System, Long Beach, California
  - San Francisco VA Health Care System", San Francisco, California
  - Lundquist Institute for Biomedical Innovation at Harbor - UCLA Medical Center, Torrance, California
  - Invivocure, Van Nuys, California
  - Interventional Cardiology Medical Group, West Hills, California
  - Colorado Heart and Vascular PC, Golden, Colorado
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Christiana Care Health Services, Inc., Newark, Delaware
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - FWD Clinical Research, Boca Raton, Florida
  - Bay Area Cardiology Associates, P.A., Brandon, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Pioneer Clinical Studies (PCS), Coral Gables, Florida
  - University of Florida Health Science Center at Jacksonville, Jacksonville, Florida
  - Baptist Health Research Institute, Jacksonville, Florida
  - Baptist Health Care, Inc. d/b/a Baptist Hospital Cardiology, Pensacola, Florida
  - Ascension Sacred Heart, Pensacola, Florida
  - Clearwater Cardiovascular Consultants, Safety Harbor, Florida
  - Centricity Research Columbus Georgia Multispecialty, Columbus, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Endeavor Health, Glenview, Illinois
  - OSF HealthCare Cardiovascular Institute, Peoria, Illinois
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Indiana University Health Ball Memorial Hospital, Muncie, Indiana
  - Reid Physician Associates, Richmond, Indiana
  - St. Elizabeth Healthcare, Edgewood, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Grace Research, LLC, Bossier City, Louisiana
  - Heart Clinic of Hammond, Hammond, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Sinai Hospital Baltimore, LifeBridge Health, Baltimore, Maryland
  - Adventist Healthcare White Oak Medical Center, Silver Spring, Maryland
  - Profound Research LLC at Millenium Cardiology, Farmington Hills, Michigan
  - MyMichigan Medical Center - Midland, Midland, Michigan
  - Regions Hospital, Saint Paul, Minnesota
  - Cardiology Associates Research, Tupelo, Mississippi
  - University of Missouri Healthcare, Columbia, Missouri
  - North Kansas City Hospital, North Kansas City, Missouri
  - Advanced Heart Care, LLC, Bridgewater, New Jersey
  - Saint Michael's Medical Center, Newark, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - AtlantiCare Regional Medical Center, Pomona, New Jersey
  - Bassett Medical Center, Cooperstown, New York
  - St. Joseph's Hospital Cardiology, Liverpool, New York
  - VA NY Harbor Healthcare System, New York, New York
  - University of Rochester - PARENT, Rochester, New York
  - Mecklenburg Heart Specialists, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Moses H. Cone Memorial Hospital Operation Corporation d/b/a Cone Health, Greensboro, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Wellspan Chambersburg Hospital, Chambersburg, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Penn State Health Medical Group - Berks Cardiology, Wyomissing, Pennsylvania
  - Prisma Health - Upstate, Greenville, South Carolina
  - Upstate Cardiology, Greenville, South Carolina
  - Monument Health Clinical Research, Monument Health Rapid City Hospital Inc., Rapid City, South Dakota
  - CHI Institute for Research and Innovation, Chattanooga, Tennessee
  - Baptist Clinical Research Institute, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Covenant Medical Group d/b/a Parkway Cardiology Associates, Oak Ridge, Tennessee
  - Cardiovascular Research of Knoxville, Powell, Tennessee
  - Amarillo Heart Clinical Research Institute Inc., Amarillo, Texas
  - PharmaTex Research, Amarillo, Texas
  - North Texas Research Associates, McKinney, Texas
  - UVA University Hospital, Charlottesville, Virginia
  - Inova Heart & Vascular Institute, Falls Church, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Bon Secours St. Mary's Hospital of Richmond, LLC, Richmond, Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Australia (14):
  - Royal Adelaide Hospital/ CNARTS, Adelaide
  - Grampians Health, Ballarat
  - The Prince Charles Hospital, Chermside
  - Monash Health, Clayton
  - Concord Repatriation General Hospital (CRGH) (Concord Hospital), Concord
  - The Cardiologists Pty. Ltd, Epping
  - The Canberra Hospital, Garran
  - Gosford Hospital, Gosford
  - Tasmanian Health at Royal Hobart Hospital, Hobart
  - The Alfred Hospital, Melbourne
  - Core Research Group Pty Ltd, Milton
  - Western Health - Sunshine Hospital, St Albans
  - Wollongong Hospital - Illawarra Shoalhaven Local Health District, Wollongong
  - The Queen Elizabeth Hospital, Woodville South
- Austria (5):
  - LKH Universitätsklinikum Graz, Graz
  - Klinikum Klagenfurt am Woerthersse, Klagenfurt
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Klinik Ottakring, Vienna
  - Karl Landsteiner Institut für Kardiovaskuläre und Intensivmedizinische Forschung, Vienna
- Belgium (5):
  - OLV Aalst, Aalst
  - Hospital Oost-Limburg (ZOL), Genk
  - AZ Sint-Lucas, Ghent
  - University Hospital Leuven (UZ Leuven), Leuven
  - AZ Delta Campus Rumbeke, Roeselare
- Brazil (18):
  - Hospital de Amor Barretos - Fundação PIO XII, Barretos
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - CARDRESEARCH - Cardiologia Assistencial e de Pesquisa, Belo Horizonte
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul
  - IPECC - Instituto de Pesquisa Clínica de Campinas, Campinas
  - Hospital Universitario Maria Aparecida Pedrossian, Campo Grande
  - Galileo Medical Research LTDA, Juiz de Fora
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - Instituto de Cardiologia do Rio Grande do Sul/ Fundação Universitária de Cardiologia, Porto Alegre
  - CoraCentro Pesquisa Clínica, Porto Alegre
  - Hospital Nossa Senhora da Conceição / FZ Cardiologia, Porto Alegre
  - Esho Empresa de Serviços Hospitalares- HOSPITAL PRÓ CARDIACO, Rio de Janeiro
  - Hospital e Maternidade Anna Nery, Salvador
  - Hospital Santa Izabel - Santa Casa de Misericórdia da Bahia, Salvador
  - Hospital Nove de Julho - Ímpar Serviços Hospitalares S.A, São Paulo
  - Instituto do Coração do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Ebserh Hospital de Clínicas da Universidade Federal de Uberlândia-HC-UFU, Uberlândia
- Bulgaria (22):
  - Mbal Puls, Blagoevgrad
  - MHAT Heart and Brain - Burgas, Burgas
  - UMHAT Deva Maria, Burgas
  - MHAT "Dr. Tota Venkova", AD, Gabrovo
  - MHAT Ivan Skenderov EOOD, Gotse Delchev
  - Medical Centre Avitzena, Kardzhali
  - MHAT Cardiolife OOD, Lovech
  - MHAT Uni Hospital, Panagyurishte
  - SHATC Sveti Georgi, Pernik
  - MHAT Heart and Brain - Pleven, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - Medical Center Sveti Ivan Rilski Chudotvorets-2010" EOOD, Plovdiv
  - UMHAT-Plovdiv AD, Plovdiv
  - MHAT "Sv. Karidad", EAD, Plovdiv
  - MHAT South-West Hospital, Cardiology Department, Sandanski
  - Second MHAT - Sofia AD, Sofia
  - MHAT "Lozenets", Sofia
  - UMHAT "Sveta Ekaterina", Sofia
  - UMHATEM N I Pirogov EAD, Sofia
  - MHAT-Medical Complex Sveti Ivan Rilski EOOD-branch Stara Zagora, Stara Zagora
  - MDHAT 'Dr. Stefan Cherkezov', AD, Veliko Tarnovo
  - MHAT "Sv. Panteleymon" - Yambol, AD, Yambol
- Canada (19):
  - University of Calgary Foothills Medical Centre, Calgary, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Wiliam Osler Health System, Brampton, Ontario
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - York PCI Group, Inc., Newmarket, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Clinique de Cardiologie de Lévis, Lévis, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - CHUM - Centre hospitalier de l'Universite de Montreal", Montreal, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal, Quebec
  - Centre Intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec, Trois-Rivières, Quebec
  - Hôpital du Sacré-Coeur de Montréal, Montreal
  - University of Ottawa Heart Institute, Ottawa
  - Diex Research, Inc., Trois-Rivières
  - St. Boniface Hospital, Winnipeg
- Chile (4):
  - Cec-Suecia, Santiago
  - Pontificia Universidad Catolica de Chile, Santiago
  - Clinica Ensenada, Santiago
  - Hospital San Jose de Victoria, Victoria
- China (95):
  - Baotou Central Hospital, Baotou
  - Beijing Anzhen Hospital, Capital Medical University, Beijing
  - Beijing Luhe Hospital, Capital Medical University, Beijing
  - Beijing Pinggu Hospital, Beijing
  - Cangzhou Central Hospital, Cangzhou
  - The First Bethune Hospital of Jilin University, Changchun
  - The Second Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - The Third Xiangya Hospital of Central South University, Changsha
  - Chengdu Second People's Hospital, Chengdu
  - West China Hospital of Sichuan University, Chengdu
  - The Second Hospital of Dalian Medical University, Dalian
  - Daqing Oilfield General hospital, Daqing
  - Sinopharm Coal General Hospital, Datong
  - Beijing Hospital, Dongcheng
  - Dongguan People's Hospital, Dongguan
  - Dongying People's Hospital, Dongying
  - Fujian Provincial Hospital, Fuzhou
  - Gaozhou People 's Hospital, Gaozhou
  - The First Affiliated Hospital of Shantou University Medical College, Guangdong
  - Guangdong Provincial People's Hospital, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Hospital, Hangzhou
  - Zhejiang provincial Peoples Hospital, Hangzhou
  - Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine, Hangzhou
  - The second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - The First Affiliated Hospital of Harbin Medical University, Harbin
  - Heilongjiang Provincial Hospital, Harbin
  - The First Affiliated Hospital of USTC(Anhui Provincial Hospital), Hefei
  - Jiaozuo People's Hospital, Jiaozuo
  - Jieyang People's Hospital, Jieyang
  - Shandong University Qilu Hospital, Jinan
  - Jinan Central Hospital, Jinan
  - The First Affiliated Hospital of Shandong First Medical University (Shandong Provincial Qianfoshan Hospital), Jinan
  - The Second Hospital of Shandong University, Jinan
  - Jining No.1 People's Hospital, Jining
  - Yan'an Hospital Affiliated to Kunming Medical University, Kunming
  - Gansu Provincial Hospital, Lanzhou
  - Lianyungang First People's Hospital, Lianyungang
  - Liaocheng people's Hospital, Liaocheng
  - Linyi People's Hospital, Linyi
  - Henan University of Science and Technology (HUST) - The First Affiliated Hospital, Luoyang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Beijing Anzhen Nanchong Hospital, Capital Medical University & Nanchong Central Hospital, Nanchong
  - Nanjing Drum Tower Hospital, Nanjing
  - Zhongda Hospital Southeast University, Nanjing
  - Nanjing Jiangning Hospital, Nanjing
  - Nanyang Central Hospital, Nanyang
  - Nanyang Second People's Hospital, Nanyang
  - The first affiliated Hospital of Ningbo University, Ningbo
  - Ningbo Medical Center Lihuili Hospital, Ningbo
  - Pingxiang People's Hospital, Pingxiang
  - Qingdao Municipal Hospital, Qingdao
  - Ruian Peoples Hospital, Rui’an
  - Shanghai Ninth People's hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Chest Hospital ,Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Tenth People 's Hospital, Shanghai
  - Shanghai General Hospital, Shanghai
  - Shanghai East Hospital (Tongji University East Hospital), Shanghai
  - Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Jiading Central Hospital, Shanghai
  - Yuebei People's Hospital, Shaoguan
  - Zhuji People's Hospital, Shaoxing
  - The fourth Affiliated Hospital of China Medical University, Shenyang
  - The People's Hospital of Liaoning Province, Shenyang
  - The first Hospital of Hebei Medical University, Shijiazhuang
  - The Third Hospital of Shijiazhuang, Shijiazhuang
  - The Second Hospital of Hebei Medical University, Shijiazhuang
  - The Fourth Affiliated Hospital of Soochow University, Suzhou
  - The first Affiliated Hospital of Soochow, Suzhou
  - Shanxi Cardiovascular Hospital, Taiyuan
  - Tangshan Central Hospital, Tangshan
  - Tianjin Medical University General Hospital, Tianjin
  - Tianjin Fourth Central Hospital, Tianjin
  - Tianjin Chest Hospital, Tianjin
  - Teda International Cardiovascular Hospital, Tianjin
  - Wenzhou Medical University (WMU) - The First Affiliated Hospital, Wenzhou
  - Wenzhou People's Hospital, Wenzhou
  - The Central Hospital of Wuhan, Wuhan
  - Wuhan Asia Heart Hospital, Wuhan
  - Renmin Hospital of Wuhan University, Wuhan
  - The People's Hospital of Wuxi, Wuxi
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First Affiliated Hospital of Xinjiang Medical University, Xinjiang
  - Xinxiang Central Hospital, Xinxiang
  - Xuzhou Medical University Affiliated Hospital, Xuzhou
  - Northern Jiangsu People's Hospital, Yangzhou
  - Yanbian University Affiliated Hospital, Yanji
  - Yiyang Central Hospital, Yiyang
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang
  - Zhanjiang Central People 's Hospital, Zhanjiang
  - The 7th People's Hospital of Zhengzhou, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou
  - Zibo Central Hospital, Zibo
- Colombia (11):
  - Cardiomet Cequin S.A.S, Armenia
  - Hospital Universitario San Ignacio, Bogotá
  - Fundación Cardioinfantil - Instituto de Cardiología, Bogotá
  - Administradora Country S.A.S. - Clinica del Country, Bogotá
  - Fundación Valle del Lili, Cali
  - IPS Centro Médico Julián Coronel S.A.S, Cali
  - Clinica Imbanaco S.A.S, Cali
  - Fundación cardiovascular de Colombia, Floridablanca
  - Hospital Alma Mater de Antioquia, Medellín
  - Rodrigo Botero SAS, Medellín
  - Clinica Cardio VID, Medellín
- Czechia (18):
  - ICRC St. Anne University Hospital, Brno
  - University Hospital Brno, Brno
  - Kardiologie Bruntál CorMedico s.r.o, Bruntál
  - Regional Hospital Ceské Budejovice, České Budějovice
  - University hospital Hradec Králové, Hradec Králové
  - Regional Hospital Jihlava, Jihlava
  - Regional Hospital Liberec, Liberec
  - KARDIOKRI s.r.o, Ostrava - Poruba
  - Nemocnice Pardubickeho kraje, a.s. - Pardubicka nemocnice, Pardubice
  - Fakultní nemocnice Plzen, Pilsen
  - Univ. Hospital Vinohrady, Prague
  - Kardiologie Praha s.r.o., Prague
  - General Faculty Hospital, Prague
  - Všeobecná fakultní nemocnice, Prague
  - Institutu Klinicke a Experimentalni Mediciny (IKEM) (Institute for Clinical and Experimental Medicine), Prague
  - Kardiologie Vinohrady s.r.o., Praha 1 - Nové Mesto
  - Olomuc Cardiology, Prostějov
  - University Hospital Ústí nad Labem, Ústí nad Labem
- Denmark (10):
  - Aalborg University Hospital Cardiology, Aalborg
  - Aarhus University Hospital, Aarhus
  - Esbjerg Hospital, Esbjerg
  - Rigshospitalet, Hellerup
  - Goedstrup Region Hospital, Herning
  - Herning Hospital, Herning
  - Odense Universitetshospital, Odense
  - Zealand University Hospital, Roskilde
  - Svendborg Hospital, Svendborg
  - Viborg Hospital, Viborg
- Estonia (2):
  - The North Estonia Medical Centre, Tallinn
  - Heart Clinic, Tartu University Hospital, Tartu
- Finland (11):
  - Jorvi Hospital, Helsinki University Hospital, Espoo
  - Heart and Lung Center, Helsinki University Hospital, Helsinki
  - North Karelian Central Hospital, Joensuu
  - StudyCor, Jyväskylä
  - Kokkola Central Hospital, Kokkola
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Seinäjoki Central Hospital, Seinäjoki
  - TAYS Tutkimusvastaanotto / TAYS Research Center, Tampere
  - TAYS Sydänkeskus Oy (Heart Hospital Tampere University Hospital), Tampere
  - Heart Center, Turku University Hospital, Turku
- France (14):
  - Hopital Cardiologique CHU Bordeaux, Pessac, Gironde
  - CHRU Brest - Cavale Blanche, Brest
  - CHU Caen · Unité Cardiologie et Pathologie Vasculaire, Caen
  - Hospital Center Departmental Vendée, La Roche-sur-Yon
  - CH Chartres, Le Coudray
  - CHU Timone 2, Marseille
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Clinique du Millénaire, Montpellier
  - Univ Hosp de Nimes Carémeau, Nîmes
  - University Hospitals Pitié Salpêtrière, Paris
  - Bichat-Claude Bernard Hospital, Paris
  - Nouvel Hopital Civil, Strasbourg
  - Hosp Rangueil - Cardiology A Dept, Toulouse
  - CHRU Nancy, Vandœuvre-lès-Nancy
- Georgia (14):
  - High Technology Hospital Medcenter, Batumi
  - LLC " Geo Hospitals", Gurjaani
  - LTD West Georgia Medical Center, Kutaisi
  - LTD"West Regional Center of the Modern Medical Technologies, Kutaisi
  - Aleksandere Aladashvili Clinic, Tbilisi
  - JSC Viani, Tbilisi
  - LLC Geo Hospitals, Tbilisi
  - Ltd Cardiology Clinic "Guli", Tbilisi
  - Acad. G. Chapidze Emergency Cardiology Center, Tbilisi
  - Bokhua Memorial CardioVascular Center, Tbilisi
  - Tbilisi Heart and Vascular Clinic Ltd., Tbilisi
  - TIM Hospital, Tbilisi
  - Georgian-Dutch hospital, Tbilisi
  - LTD "Tbilisi Heart Center", Tbilisi
- Germany (22):
  - Universitätsklinikum Freiburg; Universitäts-Herzzentrum Freiburg-Bad Krozingen, Bad Krozingen
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - MedicTRials STUG - Praxis Dr. Toursarkissian, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Krankenhaus der Augustinerinnen Köln gGmbH, Cologne
  - Universitätsklinikum Köln, Cologne
  - St. Johannes Hospital Dortmund, Dortmund
  - Herzzentrum Dresden GmbH; Universitätsklinik an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - SRH Klinikum Karlsbad-Langensteinbach GmbH, Karlsbad
  - Herzzentrum Leipzig GmbH, Leipzig
  - Gesellschaft für Klinische Forschung mbH Ludwigshafen, Ludwigshafen
  - Uniklinikum Magdeburg A. ö. R., Magdeburg
  - Universitätsmedizin Mannheim, Mannheim
  - München Klinik Neuperlach, München
  - Studienzentrum Innere Med. II Kardiologie, Universitätsklinikum Regensburg, Regensburg
  - Robert-Bosch Krankenhaus Stuttgart, Stuttgart
  - Krankenhaus der Barmherzigen Brüder, Trier
  - Universitätsklinikum Tübingen, Medizinische Klinik Innere Medizin III Kardiologie und Angiologie, Tübingen
  - Siteworks GmbH Prüfzentrum Völklingen, Völklingen
  - Helios Universitätsklinikum Wuppertal, Wuppertal
- Greece (14):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - General Hospital of Athens "Laiko", Athens
  - Ippokrateio (Hyppokration) General Hospital of Athens, Athens
  - University General Hospital "Attikon", Athens
  - University Hospital of Heraklion, Heraklion
  - Thriasio General Hospital, Magoula
  - Hygeia Hospital, Marousi
  - Sismanoglio Hospital of GNA "Sismanoglio - Amalia Fleming, Marousi
  - Konstantopouleio - Patision General Hospital of Nea Ionia, Nea Ionia
  - University Hospital of Patras, Pátrai
  - Tzaneio Hospital, Piraeus
  - Aristotle University of Thessaloniki (AUTH) - University General Hospital of Thessaloniki (AHEPA), Thessaloniki
  - General Hospital of Thessaloniki G.Papanikolaou, Thessaloniki
  - Asklepeion General Hospital, Voula, Voula
- Hungary (16):
  - Euréka-Center Bt., Baja
  - Állami Szívkorhaz, Balatonfüred
  - Betegápoló Irgalmasrend Budai Irgalmasrendi Kórház, Kardiológia, Budapest
  - Gottsegen György Országos Kardiovaszkuláris Intézet, Budapest
  - Budapesti Bajcsy-Zsilinszky Hospital, Budapest
  - Semmelweis Egyetem Városmajori Szív- és Érgyógyászati Klinika Kardiológia, Budapest
  - Magyar Honvédség Egészségügyi Központ, Budapest
  - Uzsoki Utcai Kórház, Budapest
  - Debreceni Egyetem Klinikai Központ Kardiológiai és Szívsebészeti Klinika, Debrecen
  - Bács-Kiskun Megyei Kórház a Szegedi Tudományegyetem Általános Orvostudományi Kar Oktató Kórháza, Kecskemét
  - SzSzBV Egyetemi Oktatókórház, Nyíregyházi Jósa András Tagkórház, Kardiológia, Nyíregyháza
  - Pécsi Tudományegyetem, ÁOK, Pécs
  - DaVinci Magánklinika, Pécs
  - Szegedi Tudományegyetem ÁOK Szent-Györgyi Albert Klinikai Központ II.sz. Belgyógyászati Klinika és Kardiológiai Központ, Szeged
  - Jász-Nagykun-Szolnok Megyei Hetényi Géza Kórház-Rendelőintézet, Szolnok
  - Léda-Platán Magánklinika, Zalaegerszeg
- India (51):
  - GCS Medical College, Hospital & Research Centre, Ahmedabad
  - Care Institute of Medical Sciences, Ahmedabad
  - Jawaharlal Nehru Medical College and Hospital - AMU, Aligarh
  - Kamal Nayan Bajaj Hospital, Aurangabad
  - Narayana Health - Institute of Cardiac Sciences, Bangalore
  - K.L.E. Society's Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagavi
  - BHS Lakeview Hospital, Belagavi
  - The Madras Medical Mission, Chennai
  - Sgrrih & Ms, Dehradun
  - Batra Hospital And Medical Research Centre, Delhi
  - Sarvodaya Hospital, Faridabad
  - Max Super Speciality Hospital Vaishali, Ghaziabad
  - Lalitha Super Speciality Hospital, Guntur
  - Osmania General Hospital, Hyderabad
  - Malla Reddy Narayana Multispecialty hospital, Hyderabad
  - Sri Sri Holistic Hospitals, Hyderabad
  - Apex Hospital Pvt. Ltd., Jaipur
  - SRM Medical College Hospital and Research Centre, Kattankulathur
  - Lisie Hospital, Kochi
  - Lakeshore Hospital and Research Centre Ltd., Kochi
  - Amrita Institute Of Medical Sciences and Research Centre, Kochi
  - IPGMER and SSKM Hospital, Kolkata
  - Government General Hospital, Kurnool
  - King George's Medical University, Lucknow
  - Meenakshi Mission Hospital & Research Centre, Madurai
  - Arneja Heart Institute, Nagpur
  - Crescent Hospital & Heart Centre, Nagpur
  - Central India Cardiology Hospital and Research Institute, Nagpur
  - Swasthyam Superspeciality Hospital, Nagpur
  - NKP Salve Institute of Medical Sciences, Nagpur
  - Chopda Medicare & Research Centre, Nashik
  - Vijan Cardiac and Critical Care, Nashik
  - Max Super Speciality Hospital, New Delhi
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Government Medical College and Hospital Ongole, Ongole
  - Indira Gandhi Institute of Medical Sciences, Patna
  - Moti Lal Nehru Medical College, Prayagraj
  - Sahyadri Super Speciality Hospital, Pune
  - KEM Hospital Research Center, Pune
  - Villoo Poonawalla Memorial Hospital, Pune
  - Crescent India Medical Education Trust's Inamdar Hopital, Pune
  - SMC Heart Institute and IVF Research Centre, Raipur
  - Sterling Hospital, Rajkot
  - Krishna Institute of Medical Sciences, Secunderabad
  - Nirmal Hospital Private Limited, Surat
  - Unicare Heart Institute, Surat
  - Aashirwad Hospital, Ulhasnagar
  - Rhythm Heart Institute, Vadodara
  - Government Siddhartha Medical College, Vijayawada
  - King George Hospital, Visakhapatnam
- Israel (15):
  - Soroka University Medical Center, Beersheba
  - Hillel Yaffee Medical Center, Cardiology Department, Hadera
  - Rambam Health Care Campus, Haifa
  - Bnai Zion Medical Center, Cardiology, Haifa
  - Edith Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Cardiology Department, Jerusalem
  - Hadassah Hospital on Mount Scopus, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Kaplan Medical Center, Intensive Cardiac Care Unit, Rehovot
  - Ziv Medical Center, Safed
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Leviev Heart Center, Sheba Medical Center, Tel Litwinsky
  - Shamir Medical Center (Assaf Harofeh), Ẕerifin
- Italy (15):
  - San Donato Hospital, U.O.C. Cardiology, Arezzo
  - Ospedale Maggiore Bologna - Dept. Cardiology, Bologna
  - AORN "Sant'Anna e San Sebastiano", Caserta
  - Azienda Ospedaliero-Universitaria Policlinico ""G. Rodolico - San Marco, Catania
  - Azienda Ospedaliero-Universitaria Policlinico "G. Rodolico - San Marco", Catania
  - AOU Mater Domini, Catanzaro
  - University Hospital of Ferrara, Cardiology Unit, Cona
  - "SOD Cardiologia Interventistica Strutturale, AOU Careggi, Florence
  - A.O.U. Policlinico Gaetano Martino, Messina
  - University of Naples "Federico II", Napoli
  - AOU San Luigi Gonzaga Hospital, Orbassano
  - Azienda Ospedaliera di Perugia, Perugia
  - A.O.U.Città della Salute e della Scienza di Torino, Torino
  - Cardiology Department - Santa Chiara Hospital, Trento
  - Infermi Hospital in Rivoli (Turin), Turin
- Japan (40):
  - Hyogo Prefectural Amagasaki General Medical Center, Amagasaki-shi
  - Asahi General Hospital, Asahi-shi
  - Nippon Medical School Hospital, Bunkyō City
  - Fukuokaken Saiseikai Futsukaichi Hospital, Chikushino-shi
  - Tokushukai Nozaki Tokushukai Hospital, Daito-shi
  - Chiyukai Fukuoka Wajiro Hospital, Fukuoka
  - Kenshinkai Minamino Cardiovascular Hospital, Hachioji-shi
  - Hakodate Municipal Hospital, Hakodate-shi
  - Seirei Hamamatsu General Hospital, Hamamatsu
  - Hyogo Prefectural Harima-Himeji General Medical Center, Himeji-shi
  - Hiratsuka Kyosai Hospital, Hiratsuka-shi
  - Juntendo University Shizuoka Hospital, Izunokuni-shi
  - Tokushukai Shonan Kamakura General Hospital, Kamakura-shi
  - Ibaraki Prefectural Central Hospital, Kasama-shi
  - Kasugai Municipal Hospital, Kasugai-shi
  - Kimitsu Chuo Hospital, Kisarazu-shi
  - Sakurakai Takahashi Hospital, Kobe
  - NHO Fukuoka Higashi Medical Center, Koga-shi
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Japanese Red Cross Kumamoto Hospital, Kumamoto
  - Omi Medical Center, Kusatsu-shi
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - NHO Tokyo Medical Center, Meguro-ku
  - Japanese Red Cross Musashino Hospital, Musashino-shi
  - Nagasaki Harbor Medical Center, Nagasaki
  - Japanese Red Cross Aichi Medical Center Nagoya Daini Hospital, Nagoya
  - Ome Medical Center, Ome-shi
  - NHO Nagasaki Medical Center, Omura-shi
  - NHO Osaka National Hospital, Osaka
  - Osaka General Medical Center (Kyuseiki Sogo Iryo C), Osaka
  - NHO Oita Medical Center, Ōita
  - Saga-Ken Medical Centre Koseikan, Saga
  - Kitasato University Hospital, Sagamihara-shi
  - Kosekai Iwatsuki-minami Hospital, Saitama-shi
  - Tokyo Metropolitan Hiroo Hospital, Shibuya-ku
  - Mie University Hospital, Tsu
  - Yamaguchi University Hospital, Ube-shi
  - Tokyobay Urayasu Ichikawa Medical Center, Urayasu-shi
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama
  - Yokohama Sakae Kyosai Hospital, Yokohama
- Lithuania (4):
  - Hospital of Lithuanian University of Health Sciences Kauno Klinikos, Kaunas
  - Klaipeda Seamen's Hospital, Klaipėda
  - Republican Panevezys Hospital, Panevezys
  - Vilnius University Hospital Santaros Klinikos, Vilnius
- Mexico (9):
  - Hospital Cardiológica Aguascalientes, Aguascalientes
  - Centro para el desarrollo de la medicina y de asistencia médica especializada S.C., Culiacán
  - Boca Clinical Trials México, SC (CDMX), Mexico City
  - Instituto Nacional de Cardiología "Ignacio Chávez", Mexico City
  - Fundación de Atención e Investigación Médica Lindavista S.C, Mexico City
  - Boca Clinical Trials México, SC (Puebla), Puebla City
  - SMIQ / Boca Clinical Trials México, Querétaro
  - Centro de Atención e Investigación Cardiovascular del Potosí, S.C., San Luis Potosí City
  - Centro Potosino de Investigación Médica S.C., San Luis Potosí City
- Netherlands (22):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Meander Medisch Centrum, Amersfoort
  - Onze Lieve Vrouwe Gasthuis, locatie Oost, Amsterdam
  - Amsterdam UMC, Amsterdam
  - Gelre Ziekenhuis Apeldoorn, Apeldoorn
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Gelderse Vallei Ziekenhuis, Ede
  - Catharina Hospital, Eindhoven
  - Admiraal de Ruyter Ziekenhuis, Goes
  - UMC Groningen, Groningen
  - Zuyderland Medical Center, Heerlen
  - Vasculair Onderzoek Centrum Hoorn, Hoorn
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Radboud UMC, Nijmegen
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Bravis Ziekenhuis, Roosendaal
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Diakonessenhuis Utrecht, Utrecht
  - Máxima Medisch Centrum, Veldhoven
- New Zealand (4):
  - Waikato Hospital, Hamilton
  - Taranaki Base Hospital, New Plymouth
  - Health New Zealand Te Whatu Ora Lakes, Rotorua
  - Bay of Plenty Clinical School Charitable Trust, Tauranga
- Norway (10):
  - Sørlandet Hospital Arendal, Arendal
  - Ålesund Hospital, Ålesund
  - Nordland Hospital Trust, Bodø
  - Akershus University Hospital, Lørenskog
  - Diakonhjemmet Hospital, Oslo
  - Oslo University Hospital Rikshospitalet, Oslo
  - Oslo University Hospital, Ullevål hospital, Oslo
  - Sykehuset Østfold Kalnes (Trust), Sarpsborg
  - Stavanger University Hospital, Stavanger
  - Vestfold Hospital, Tønsberg
- Poland (24):
  - Invasive Cardiology Department, University Teaching Hospital in Białystok, Bialystok
  - Specjalistyczna Praktyka Lekarska Paweł Grzelakowski Centrum Kardiologii Paewł Grzelakowski, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Clinical Medical Research Sp. z o.o., Katowice
  - Gyncentrum Sp. z o.o., Katowice
  - Górnośląskie Centrum Medyczne w Katowicach, III Oddział Kardiologii, Katowice
  - Szpital Uniwersytecki w Krakowie, Oddział Kliniczny Kardiologii oraz Interwencji Sercowo-Naczyniowych, Krakow
  - Linden Sp. z o.o. sp.k., Krakow
  - Nzoz Salusmed Jan Zbigniew Peruga Pphu Salus Poradnia Kardiologiczna, Lodz
  - Centrum Medyczne Med-GASTR SP. Z O.O, Lodz
  - Wojewodzki Szpital Specj im.W Bieganskiego, LÓDZ
  - Zanamed Medical Clinic sp z o o, Lublin
  - Miedziowe Centrum Zdrowia Regionalny, Ośrodek Kardiologiczny, Pracownia Angiografii i Hemodynamiki, Lublin
  - Wojewódzki Szpital Specjalistyczny w Olsztynie, Oddział Kardiologii, Olsztyn
  - INKARD Sp. Z O.O. Sp. JAWNA, Poznan
  - Szpital Kliniczny im. Heliodora Swiecickiego Uniwersytetu Medycznego im. Karola Marcinkowskiego w Poznaniu, Poznan
  - Wojewodzki Szpital im. Sw. Ojca Pio w Przemyslu, Przemyśl
  - Oddzial Kardiologii i intensywnej Terapii Kardiologicznej, Torun
  - Pracownia Kardiologii Inwazyjnej I Katedry i Kliniki Kardiologii Uniwersyteckiego Centrum Klinicznego Warszawskiego Uniwersytetu Medycznego, Warsaw
  - Narodowy Instytut Kardiologii, Warsaw
  - Uniwersytecki Szpital Kliniczny we Wroclawiu, Wroclaw
  - Dolnoslaski Szpital Specjalistyczny im. T.Marciniaka - Centrum Medycyny Ratunkowej, Wroclaw
  - The Provincial Specialist Hospital in Wloclawek, Włocławek
  - SCCS Zabrze I i II Oddział Kardiologii i Angiologii, Zabrze
- Portugal (5):
  - Unidade Local de Saúde de Almada-Seixal, E.P.E., Almada
  - Unidade Local de Saúde da Região de Aveiro, E.P.E., Aveiro
  - Unidade Local de Saude de Coimbra EPE, Coimbra
  - Unidade Local de Saúde da Região de Leiria, E.P.E., Leiria
  - Unidade Local de Saúde de Santa Maria, E.P.E., Lisbon
- Romania (16):
  - Spitalul Judetean de Urgenta ""Dr. Constantin Opris" Baia Mare, Baia Mare
  - Spitalul Judetean de Urgenta "Dr. Constantin Opris" Baia Mare, Baia Mare
  - Centrul Medical Unirea S.R.L, Brasov
  - County Clinical Emergency Hospital Brasov, Brasov
  - Spitalul Clinic de Urgenta Bucuresti, Bucharest
  - Spitalul Universitar de Urgenta Militar Central "Dr. Carol Davila", Bucharest
  - Delta Health Care SRL, Bucharest
  - Institutul Inimii de Urgență pentru Boli Cardiovasculare "Niculae Stăncioiu", Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic Judetean de Urgenta Craiova, Craiova
  - Spitalul Clinic Judetean De Urgenta Bihor, Oradea
  - Spitalul Judetean de Urgenta Satu Mare, Satu Mare
  - County Clinical Emergency Hospital Targu Mures, Târgu Mureş
  - Podoleanu G. Cristian-Gheorghe-Calin - Cabinet Medical De Cardiologie, Târgu Mureş
  - Spitalul Clinic Municipal de Urgenta Timisoara, Timișoara
  - Institute of Cardiovascular Diseases Timisoara, Timișoara
- Serbia (17):
  - Kliničko bolnički centar "Zvezdara", Belgrade
  - University Clinical Center of Serbia (Department for Cardiovascular Disease Cardiology Clinic), Belgrade
  - University Clinical Center of Serbia (Diagnostic and Catheterization Lab), Belgrade
  - University Clinical Center of Serbia (Emergency Cardiology Services), Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Hospital Centre Dr Dragiša Mišovic - Dedinje, Belgrade
  - Dedinje Cardiovascular Institute, Belgrade
  - Clin Hosp Ctr Zemun - Cardiology Dept, Belgrade
  - Department of Cardiology, Clinical Hospital Center Zemun, Belgrade
  - Klinicko bolnicki centar, Bežanijska kosa, Belgrade
  - Kliničko Bolnički Centar Bežanijska Kosa, Belgrade
  - Institute of Cardiovascular Diseases, Vojvodina, Kamenitz
  - Klinički centar Kragujevac, Kragujevac
  - Opšta bolnica Leskovac, Leskovac
  - Klinički Centar Niš, Niš
  - Opšta bolnica Užice, Užice
  - Zdravstveni Centar Zajecar, Zaječar
- Slovakia (6):
  - Central Slovak Institute of Cardiovascular Diseases, Banská Bystrica
  - Premedix Clinic, Bratislava
  - University Hospital Bratislava, Bratislava
  - Cardiocentre CINRE, Bratislava
  - Východoslovenský ústav srdcových a cievnych chorôb, Košice
  - Kardiocentrum Nitra, Nitra
- South Africa (7):
  - Iatros International, Bloemfontein
  - Josha Research, Bloemfontein
  - Tread Research, Cape Town
  - Synergy Biomed Research Institute (SBRI), East London
  - Futurex Clinical, Johannesburg
  - Eden Heart, Mossel Bay
  - Paarl Research Centre, Paarl
- South Korea (13):
  - The Catholic University of Korea, Bucheon, St. Mary's Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Ewha Womans University Seoul Hospital, Gangseo-gu
  - Myongji Hospital, Goyang-si
  - Gachon University Gil Medical Center, Incheon
  - Kyung Hee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul
  - Asan Medical Center, Seoul
- Spain (11):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital Clinic. Barcelona, Barcelona
  - Hospital Universitario Virgen de la Arrixaca, El Palmar
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Clinico Valencia, Valencia
  - Hospital Alvaro Cunqueiro, Cardiovascular Unit, Vigo
- Switzerland (4):
  - Universitätsspital Basel; Universitäres Herzzentrum, Basel
  - Inselspital, Universitäatspital Bern, Universitäatklinik für Kardiologie, Bern
  - Istituto Cardiocentro Ticino, Lugano
  - HOCH Health Ostschweiz, Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (13):
  - Changhua Christian Hospital, Changhua
  - Hualien Tzu Chi Hospital, Hualien City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chang Gung Medical Foundation-Kaohsiung, Kaohsiung City
  - Mackay Memorial Hospital Tamsui, New Taipei City
  - Chung Shan Medical University Hospital, Taichung, Taichung
  - Chi Mei Medical Center, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - TRI-Service General Hospital, Taipei
  - Taitung MacKay Memorial Hospital, Taitung
  - Linkou Chang Gung Memorial Hospital, Taoyuan
- Thailand (9):
  - Bhumibol Adulyadej Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Faculty of Medicine, Chiang Mai University, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Chiang Rai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Thammasat University Hospital, Pathum Thani
  - Buddhachinaraj Phitsanulok Hospital, Phitsanulok
  - Songklanagarind Hospital, Songkhla
  - Fort Sanpasitthiprasong Hospital, Ubon Ratchathani
- United Kingdom (9):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - Barts Health NHS Trust, London
  - Altnagelvin Area Hospital (WHSCT), Londonderry
  - Freeman Hospital, Newcastle
  - North Tyneside General Hospital, Northumbria Healthcare, North Shields
  - Southern Health & Social Care Trust, Portadown
  - Northern General Hospital, Sheffield
  - Lister Hospital East and North Hertfordshire NHS Trust, Stevenage
  - Worcestershire Acute Hospital NHS Trust, Worcester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thygesen K, Alpert JS, Jaffe AS, Chaitman BR, Bax JJ, Morrow DA, White HD; Executive Group on behalf of the Joint European Society of Cardiology (ESC)/American College of Cardiology (ACC)/American Heart Association (AHA)/World Heart Federation (WHF) Task Force for the Universal Definition of Myocardial Infarction. Fourth Universal Definition of Myocardial Infarction (2018). J Am Coll Cardiol. 2018 Oct 30;72(18):2231-2264. doi: 10.1016/j.jacc.2018.08.1038. Epub 2018 Aug 25. No abstract available. PMID 30153967
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242